CLINICAL TRIAL: NCT02983253
Title: Immunmodulation in Patients With HHT
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Urban Geisthoff, Prof. Dr. med. Urban Geisthoff, University Hospital, Essen
Other Study IDs: ImmunUHEssen
Record Dates: First submitted 2016-12-02; First posted 2016-12-06 (Estimated); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Hereditary Haemorrhagic Telangiectasia (HHT)
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with HHT: blood sample of patients with HHT
  Interventions: Other: blood sample
- probands: blood sample of healthy controls
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — none, only laboratory tests on blood serum

SUMMARY:
Hereditary haemorrhagic telangiectasia (HHT), also known as Rendu-Osler-Weber syndrome, is an inherited multisystemic disorder. Literature suggests that HHT is often associated with higher frequency of infectious diseases.

The purpose of this study is to evaluate a variety of immunologic parameters in the blood serum of HHT patients in comparison to probands.

DETAILED DESCRIPTION:
Hereditary haemorrhagic telangiectasia (HHT), also known as Rendu-Osler-Weber syndrome, is an inherited multisystemic disorder with recurrent epistaxis, mucocutaneous telangiectasia and visceral arteriovenous malformations. Literature and the investigators' observation suggest that HHT is often associated with higher frequency of infectious diseases. This might be a hint for a immunocompromised situation.

The purpose of this study is to evaluate a variety of immunologic parameters in the blood serum of HHT patients in comparison to probands.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over, HHT

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria: Aged 18 or over, HHT,
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2016-06; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Amounts of leucocytes in patients with HHT | November 2016 - December 2018

SECONDARY OUTCOMES:
Differences in distribution of leucocytes in patients with HHT | November 2016 - December 2018

OTHER OUTCOMES:
Functional properties of leucocytes in patients with HHT | November 2016 - December 2018
Differences in size of leucocytes in patients with HHT | November 2016 - December 2018

CONTACTS AND LOCATIONS:
Overall Officials: Urban Geisthoff, Prof.Dr.med., Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Undecided